CLINICAL TRIAL: NCT00119301
Title: Phase I Study of High Dose Methotrexate With Simultaneous Trimetrexate and Leucovorin in Patients With Recurrent Osteosarcoma
Brief Title: Methotrexate, Trimetrexate Glucuronate, and Leucovorin in Treating Patients With Refractory or Recurrent Osteosarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 05-028; MSKCC-IRB-05028
Record Dates: First submitted 2005-07-12; First posted 2005-07-13 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Sarcoma
Keywords: recurrent osteosarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma | interventions — Leucovorin; Methotrexate; trimetrexate glucuronate

INTERVENTIONS:
Drug: leucovorin calcium
Drug: methotrexate
Drug: trimetrexate glucuronate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as methotrexate, trimetrexate glucuronate, and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of trimetrexate glucuronate when given together with methotrexate and leucovorin in treating patients with refractory or recurrent osteosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of trimetrexate glucuronate when administered with high-dose methotrexate and leucovorin calcium in patients with refractory or recurrent high-grade osteosarcoma.

Secondary

* Determine the dose-limiting toxic effects of this regimen in these patients.
* Determine, preliminarily, the antitumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of trimetrexate glucuronate.

Patients receive high-dose methotrexate IV over 4 hours on days 1 and 8 and oral trimetrexate glucuronate twice daily on days 2-6 and 9-13. Patients also receive leucovorin calcium IV continuously over 24 hours or orally 2 or 4 times daily on days 9-14. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of trimetrexate glucuronate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A maximum of 18 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant osteosarcoma

  * High-grade disease
* Recurrent or refractory disease after prior standard chemotherapy comprising methotrexate, doxorubicin, cisplatin, and ifosfamide
* No low-grade osteosarcoma
* No parosteal or periosteal sarcoma
* No osteosarcoma arising in premalignant bony lesions (e.g., Paget's disease) OR in a prior radiotherapy field
* No symptomatic or known brain or leptomeningeal involvement

PATIENT CHARACTERISTICS:

Age

* 1 to 35

Performance status

* Karnofsky 70-100% (for patients > 16 years of age)
* Lansky 70-100% (for patients ≤ 16 years of age)

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times normal
* AST and ALT ≤ 5 times normal
* Albumin ≥ 2 g/dL
* No clinically significant liver disease

Renal

* Creatinine ≤ 1.5 times normal OR
* Creatinine clearance or radioisotope glomerular filtration rate ≥ lower limit of normal

Cardiovascular

* Shortening fraction ≥ 27% by echocardiogram OR
* Ejection fraction ≥ 50% by gated radionuclide study
* No congestive heart failure
* No angina pectoris
* No myocardial infarction within the past year
* No uncontrolled arterial hypertension
* No uncontrolled arrhythmias

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of significant neurological or psychiatric disorder
* No active infection
* No symptomatic peripheral neuropathy ≥ grade 2
* No other serious illness or medical condition

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 7 days since prior biologic therapy
* At least 6 months since prior allogeneic stem cell transplantation AND no evidence of active graft-versus-host disease
* No concurrent sargramostim (GM-CSF)

Chemotherapy

* See Disease Characteristics
* More than 2 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas)

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 6 months since prior craniospinal radiotherapy
* At least 6 months since prior radiotherapy to ≥ 50% of the pelvis
* At least 6 weeks since prior substantial radiotherapy to the bone marrow

Surgery

* Not specified

Other

* Recovered from prior therapy
* More than 30 days since prior and no other concurrent investigational drugs
* More than 30 days since prior and no concurrent participation in another clinical trial
* No concurrent medications that may interact with study drugs

Ages: 1 Year to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2005-04; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) after 1 course of treatment
Dose-limiting toxicities as assessed by hematology and biochemistry testing on days 1, 8, and 28 of each course

SECONDARY OUTCOMES:
Antitumor activity as measured by radiographic response using RECIST criteria after every 2 courses of treatment
Antitumor activity as measured by pathologic response using the Huvos grading system to evaluate post-treatment tumor necrosis at time of tumor resection after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Meyers, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States